CLINICAL TRIAL: NCT05870371
Title: The Effectiveness of the Feldenkrais Method in Reducing Pain and Improving Functionality in Patients With Chronic Neck Pain
Brief Title: The Effect of the Feldenkrais Method on Pain and Function in Patients With Chronic Neck Pain
Acronym: FMvsCNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Skordis Charalampos, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103276/18-12-2020; Research and Ethics Committee (Registry Identifier: Medical School - Aretaio Hospital, NKUA, Greece)
Record Dates: First submitted 2022-09-12; First posted 2023-05-23 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
Keywords: Feldenkrais; Awareness Through Movement; Functionality; Non specific; Chronic Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feldenkrais Awareness Through Movement (Experimental): Application of the Feldenkrais Awareness Through Movement technique in group sessions.
  Interventions: Behavioral: Feldenkrais Awareness Through Movement technique
- Acupuncture and Stretching (Active Comparator): Acupuncture protocol in combination with stretching exercises.
  Interventions: Behavioral: Acupuncture; Behavioral: Stretching

INTERVENTIONS:
Behavioral: Feldenkrais Awareness Through Movement technique — 10 group sessions, 50 minutes each, over a period of five weeks, which will include the application of the Feldenkrais Awareness Through Movement technique
  Arms: Feldenkrais Awareness Through Movement
Behavioral: Acupuncture — 10 sessions, two per week, of 25 minutes acupuncture each, which will include the insertion of a sterile disposable needle into standardized local, regional, and systematic or general acupuncture points that modify pain behavior in area of Cervical Spine.
  Arms: Acupuncture and Stretching
Behavioral: Stretching — 10 sessions, two per week, of 15 minutes stretching each, which will include lateral flexion and counterrotation of the head performed for the upper part of the trapezius and the anterior scalene, lateral flexion and corresponding rotation for the levator scapulae, and flexion for the extensors of the Cervical Spine. The following muscles will be applied: upper trapezius, levator scapulae, scalenes, extensors of the Cervical Spine (splenoid, spinous, semispinalis, longus cephalic and cervical, iliocostalis cervical, multifidus and subscapularis), and sternocleidomastoid.
  Arms: Acupuncture and Stretching

SUMMARY:
This doctoral thesis is a single blind randomized controlled clinical trial with an active control element. The intervention examined in this trial is the Awareness Through Movement (ATM) technique of the Feldenkrais Method (FM), while the standard treatment given to the control group is the combination of acupuncture and stretching.

The study was designed to examine the extend of the effect of ATM, as a means of reduction of pain, improvement of functionality and psychosomatic parameters of patients with chronic neck pain, in comparison to biomedical acupuncture protocol in combination with stretching.

The effectiveness of the intervention will be compared to the effect of the standard treatment, a combination of acupuncture and stretching, in relation to parameters of pain, range of motion of rotation, flexion-extension and lateral flexion of the cervical spine and the sense of position (kinesthesia), the endurance of the cervical deep flexor muscles, respiratory function and psychometric characteristics, which are evaluated at specific times (before and after the intervention-five weeks).

During the discussion, the results of this study, in combination with the degree of validity of the observation, will be compared to those of the literature review. This comparison could contribute to the more effective clinical application of ATM in the treatment of chronic neck pain, either as part of physiotherapeutic rehabilitation, or as a unique approach.

DETAILED DESCRIPTION:
Chronic neck pain is a common phenomenon in the adult population with a prevalence of about 15%, while it is indicative that 2/3 of the population will develop neck pain during their lifetime with slight predominance in women. In physiotherapy, a number of therapeutic techniques are available to treat chronic neck pain. Although no obvious, single treatment option has been shown to be the most effective, systematic reviews show that rehabilitation in a variety of forms has the strongest evidence for the effectiveness of relieving chronic neck pain. In these forms, complementary therapies such as acupuncture, chiropractic, yoga, Tai Chi as well as sensory-motor approaches such as the Feldenkrais method are incorporated.

Contemporary articles, found in 6 studies, investigate the effect of the Feldenkrais method (Feldenkrais Method/FM) in chronic neck pain and date between the years 1999-2014. Primary outcome measure was pain, while secondary assessed disability, functional status and quality of life. The findings in the majority showed initial positive indications for the application of FM in the management of chronic neck pain. However, further high-quality methodological studies are required in order to draw reliable conclusions.

This doctoral thesis is a single blind randomized controlled clinical trial with an active control element, where the intervention is the Feldenkrais Awareness Through Movement (ATM) technique and the standard treatment given to the control group is the combination of acupuncture and stretching, due to its scientifically proven efficacy and widespread use as the treatment of choice in this pathology.

The study was designed to examine whether and to what extent ATM application will reduce pain, improve functionality in patients with chronic neck pain and have a positive effect on the psychosomatic parameters of pain, firstly as an individual intervention and in comparison with biomedical acupuncture protocol in combination with stretching secondly.

The purpose of the study is twofold:

i. The highlight of indications for statistically significant differences in the mean values of the variables, which investigate the pain pressure threshold and objective evaluation of pain (Short Form of McGill Pain Questionnaire/SFMPQ), functionality (Neck Disability Index/NDI), range of motion of rotation, flexion-extension and lateral flexion of the cervical spine and the sense of position (kinesthesia) (3D sensor inertial motion MOOVER), the endurance of the cervical deep flexor muscles (biofeedback stabilizer pressure / Chattanooga Stabilizer Biofeedback), assessment of respiratory function (portable spirometer by MIR / MIR Spirodoc), and psychometric characteristics (Hospital Anxiety and Depression Scale/HADs, Tampa Kinesiophobia Scale/TSK_GR, SF-12 Health Survey/SF-12, Fear-Avoidance Beliefs Questionnaire/FABQ_GR, Pain Catastrophizing Scale/PCS) for group A-FM (Intervention Group-IG) and group B-acupuncture with stretching (Control Group-CG).The measurements will be performed before (pre) and after (post) of the application of the ATM technique in order to evaluate the effectiveness of each intervention separately.

ii. The comparison between the two groups, the determination of the values of the above variables before and after, during the time period of five weeks in which the two programs will be implemented in parallel.

The sample will consist of 160 patients of both sexes, aged 19-70 years, with diagnosed chronic non-specific neck pain, with a duration of pain at least three months before the initial assessment and participation in the study. The selection will be made by the method of random sampling within a period of time and the participants will be distributed by simple randomization (equal allocation) in two equal groups of 80 people each. To achieve the objectives of the study, 10 sessions will be conducted over a period of five weeks, either of the ATM technique (intervention group), lasting 50 minutes, or of biomedical acupuncture in combination with stretching (control group), 40 minutes (25 minutes acupuncture plus 15 minutes stretching). The intensity of the pain will be assessed with an algometer, the range of motion of the flexion-extension, rotation and lateral flexion and the sense of the position of the neck with 3D sensor inertial motion MOOVER, the endurance of the deep neck flexor muscles with a biofeedback stabilizer and the respiratory function with a spirometer. In addition, the sample will complete a series of questionnaires that elicit information about chronic neck pain and the dysfunction caused by chronic neck pain.

The statistical analysis will be performed with the International Business Machines (IBM) Corporation software.

The effectiveness or not of the FM will be highlighted and comparisons will be made between its effect and acupuncture plus stretching in relation to specific parameters that are evaluated at specific times (before and after the intervention-five weeks).

During the discussion, the results of this study will be compared with those of the literature review. In combination with the degree of validity of the observation (power analysis) of this study, the literature data will be taken into account and those results will be extracted, which could contribute to the more effective clinical application of FM in the treatment of chronic neck pain either as part of physiotherapeutic rehabilitation or as a unique approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic non-specific neck pain
* The duration of the symptoms should be at least three months before the initial evaluation and their participation in the study.
* Existence of reported symptoms of non-rheumatic etiology on the shoulder or upper extremity.
* Age range 19-70 years.

Exclusion Criteria:

* History of surgery in Cervical Spine (Dibai-Fihlo et al. 2017)
* Patients with a history of neck fracture or injury (Campa-Moran et al. 2015, Dibai-Fihlo et al. 2017) in the last year
* Surgery on the head, face or neck (Dibai-Fihlo et al. 2017)
* Active cervical hernia with radical symptoms or severe degenerative diseases in Cervical Spine (Dibai-Fihlo et al. 2017)
* Systemic diseases (diagnosed rheumatic, metabolic and immune diseases), (Edward & Knowles 2003, Wilke et al. 2014, Campa-Moran et al. 2015, Cerezo-Téllez et al. 2016 Dibai-Fihlo et al. 2017, Cerezo -Téllez et al. 2018)
* Myelopathy with severe disc or bone damage (Ma et al., 2010, Campa-Moran et al. 2015)
* Cervical rhizitis / rhizopathy (Ma et al. 2010, Wilke et al. 2014, Campa-Moran et al. 2015)
* Arterial dysfunction (Kerry et al. 2008)
* Tumors active during the last five years
* Lymphadenopathy (Tsakitzidis et al. 2013)
* History of inflammatory arthritis (Tsakitzidis et al. 2013)
* Diagnosed psychiatric illness (Wilke et al. 2014, Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018)
* Severe neurological disorder (Edward & Knowles 2003, Wilke et al. 2014) or mental retardation (Ma et al. 2010)
* Signs, Symptoms or History of Mouth Pain and Temporomandibular Disorders Based on the Research Diagnostic Criteria of Temporomandibular Disorders (RDC / TMD) (Campa-Moran et al. 2015)
* Fibromyalgia syndrome diagnosed (Ma et al. 2010, Wilke et al. 2014, Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018) Infection or inflammatory swelling in the treated area
* Skin damage (Edwards & Knowles 2003) or wounds in the area of the piercing (Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018)
* Systematic intake of medications that may affect the patient's judgment (eg neuromodulators, antidepressants)
* Taking systemic treatment for the same problem (Wilke et al. 2014) up to three months before the study
* Pregnancy (Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018)
* Previous Adverse Acupuncture Reaction (Edwards & Knowles 2003)
* Allergy to metal (Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018)
* Fear of the needle (Edwards & Knowles 2003, Campa-Moran et al. 2015, Cerezo-Téllez et al. 2016, Cerezo-Téllez et al. 2018)
* Inability to express speech and writing in the Greek language

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CHARALAMPOS SKORDIS, Principal Investigator — University of West Attica
Locations (2):
- Greece (2):
  - Aretaio Hospital, Athens, Attica
  - Laboratory of Musculoskeletal Physiotherapy, University of West Attica, Athens, Attica

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The physicians of the pain clinic of the 1st Anesthesiology Clinic of the Aretaeio hospital will evaluate the exclusion criteria for all patients who visit the outpatient clinics and are diagnosed with non-specific neck pain beginning on July 25, 2022, and continuing until the necessary number of participants is reached in accordance with the protocol.The patient will be assessed based on their diagnosis and exclusion criteria in order to participate in the study.
Period: Overall Study
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Started | 100 | 100
Completed | 76 | 76
Not Completed | 24 | 24
Not completed — Nonadherence (missed appointmetns). | 24 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 19-29 | 3 | 5 | 8
  Age Group: 30-39 | 6 | 13 | 19
  Age Group: 40-49 | 16 | 23 | 39
  Age Group: 50-59 | 37 | 23 | 60
  Age Group: 60-70 | 14 | 12 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 44 | 99
  Male | 21 | 32 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (5.2) | 27.5 (5.2) | 27.8 (5.2)
Education Status [Count of Participants; unit: Participants]
  None of the Below | 0 | 1 | 1
  Primary School Graduate | 6 | 1 | 7
  Secondary School Graduate | 20 | 11 | 31
  Post-Secondary Graduate | 16 | 15 | 31
  University Graduate | 28 | 37 | 65
  Post Graduate and Above | 6 | 11 | 17
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 10 | 6 | 16
  Public Sector Employment | 22 | 21 | 43
  Private Sector Employment | 25 | 39 | 64
  Self-Employed | 7 | 1 | 8
  Retirement | 12 | 9 | 21
Marital Status [Count of Participants; unit: Participants]
  Single | 14 | 13 | 27
  Married | 52 | 57 | 109
  Divorced | 8 | 6 | 14
  Windowed | 2 | 0 | 2
Symptom Duration (months) [Count of Participants; unit: Participants]
  3-6 | 6 | 8 | 14
  6-12 | 5 | 5 | 10
  12-24 | 11 | 8 | 19
  >24 | 54 | 55 | 109
Prescribed Medication Use [Count of Participants; unit: Participants]
  Yes | 30 | 21 | 51
  No | 46 | 55 | 101
Other Diseases [Count of Participants; unit: Participants]
  Yes | 38 | 36 | 74
  No | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Pain Pressure Threshold Measured by the Commander Algometer, JTECH Medical, Midvale, Utah.
Description: The selected algometer (Commander Algometer, JTECH Medical, Midvale, Utah) was used to measure pain sensitivity through the application of pressure. This device can identify the pressure eliciting a pressure-pain threshold. The pain sensitivity recording was performed at specific points with 3 measurements taken at each. The first measurement was considered tentative and was rejected and the final value was the result from the average of the two remaining measurements. The sites that were selected for the pain pressure threshold measurements were the Mastoid Process, the Bladder 10 (BL 10), the C5-C6 Zygapophyseal Joint, the Upper Trapezius Muscle, the Levator Scapula Muscle, the Deltoid Muscle and the Tibialis Anterior Muscle, bilaterally (left and right).
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: kg/cm^2
Groups:
- Acupuncture and Stretching: Acupuncture protocol in combination with stretching exercises.
  Acupuncture: 10 sessions, two per week, of 25 minutes acupuncture each, which will include the insertion of a sterile disposable needle into standardized local, regional, and general acupuncture points that modify pain behavior in area of Cervical Spine.
  Stretching: 10 sessions, two per week, of 15 minutes stretching each, which will include lateral flexion and counterrotation of the head performed for the upper part of the trapezius and the anterior scalene, lateral flexion and corresponding rotation for the levator scapulae and flexion for the extensors of the Cervical Spine. The following muscles will be applied: upper trapezius, levator scapulae, scalene, sternocleidomastoid, cervical extensor muscles (splenius, spinalis, semispinalis, longissimus capitis and cervicis and iliocostalis cervicis, multifidi and suboccipital).
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
kg/cm^2
  Mastoid Process Left (Baseline) | 1.24 (0.53) | 1.32 (0.47)
  Mastoid Process Left (Endline) | 1.61 (0.63) | 1.34 (0.51)
  Mastoid Process Right (Baseline) | 1.32 (0.52) | 1.31 (0.43)
  Mastoid Process Right (Endline) | 1.6 (0.57) | 1.32 (0.51)
  Bladder 10 Left (Baseline) | 1.76 (0.87) | 1.75 (0.52)
  Bladder 10 Left (Endline) | 2.08 (0.65) | 1.79 (0.62)
  Bladder 10 Right (Baseline) | 1.85 (0.52) | 1.85 (0.58)
  Bladder 10 Right (Endline) | 2.24 (0.66) | 1.86 (0.51)
  Zygoapophyseal Joint Left (Baseline) | 1.91 (0.58) | 1.9 (0.56)
  Zygoapophyseal Joint Left (Endline) | 2.46 (0.77) | 2.12 (0.6)
  Zygoapophyseal Joint Right (Baseline) | 1.79 (0.52) | 1.83 (0.56)
  Zygoapophyseal Joint Right (Endline) | 2.36 (0.72) | 2.12 (0.6)
  Upper Trapezius Muscle Left (Baseline) | 1.84 (0.64) | 1.74 (0.6)
  Upper Trapezius Muscle Left (Endline) | 2.2 (0.74) | 1.85 (0.68)
  Upper Trapezius Muscle Right (Baseline) | 1.95 (0.76) | 1.79 (0.73)
  Upper Trapezius Muscle Right (Endline) | 2.25 (0.83) | 2.01 (0.78)
  Levator Scapulae Muscle Left (Baseline) | 2.58 (0.84) | 2.56 (0.86)
  Levator Scapulae Muscle Left (Endline) | 3.25 (0.99) | 2.59 (0.8)
  Levator Scapulae Muscle Right (Baseline) | 2.59 (0.94) | 2.66 (0.89)
  Levator Scapulae Muscle Right (Endline) | 3.21 (1.08) | 2.84 (1.02)
  Deltoid Muscle Left (Baseline) | 2.2 (0.87) | 2.29 (0.87)
  Deltoid Muscle Left (Endline) | 2.71 (1.01) | 2.39 (0.77)
  Deltoid Muscle Right (Baseline) | 2.44 (0.93) | 2.48 (0.94)
  Deltoid Muscle Right (Endline) | 2.85 (0.83) | 2.5 (0.73)
  Tibialis Anterior Muscle Left (Baseline) | 3.24 (1.02) | 3.87 (1.3)
  Tibialis Anterior Muscle Left (Endline) | 3.83 (1.25) | 3.97 (1.59)
  Tibialis Anterior Muscle Right (Baseline) | 3.31 (1.04) | 3.85 (1.21)
  Tibialis Anterior Muscle Right (Endline) | 4.04 (1.18) | 3.95 (1.5)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null hypothesis: The application of ATM does not affect the pain sensitivity assessed by the Pain Pressure Threshold (PPT) measured with the pressure algometer (Commander Algometer) in patients with chronic neck pain (main hypothesis); Test type: Other; p = 0.002, Mixed Models Analysis — The above p value corresponds to the Mastoid Process left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.37 — The above value corresponds to the Mastoid Process left algometric site
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.018, Mixed Models Analysis — The above p value corresponds to the Mastoid Process right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.28 — The above value corresponds to the Mastoid Process right algometric site
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.020, Mixed Models Analysis — The above p value corresponds to the Bladder 10 left (BL 10) algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.32 — The above value corresponds to the Bladder 10 left (BL 10) algometric site
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.025, Mixed Models Analysis — The above p value corresponds to the Bladder 10 right (BL 10) algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.39 — The above value corresponds to the Bladder 10 right (BL 10) algometric site
Statistical Analysis 5: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p value corresponds to the Zygapophyseal Joint left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.55 — The above value corresponds to the Zygapophyseal Joint left algometric site
Statistical Analysis 6: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p value corresponds to the Zygapophyseal Joint right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.57 — The above value corresponds to the Zygapophyseal Joint right algometric site
Statistical Analysis 7: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.139, Mixed Models Analysis — The above p value corresponds to the Upper Trapezius Muscle left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.36 — The above value corresponds to the Upper Trapezius Muscle left algometric site
Statistical Analysis 8: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.011, Mixed Models Analysis — The above p value corresponds to the Upper Trapezius Muscle right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.30 — The above value corresponds to the Upper Trapezius Muscle right algometric site
Statistical Analysis 9: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.010, Mixed Models Analysis — The above p value corresponds to the Levator Scapulae Muscle left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.67 — The above value corresponds to the Levator Scapulae Muscle left algometric site
Statistical Analysis 10: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.06, Mixed Models Analysis — The above p value corresponds to the Levator Scapulae Muscle right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.62 — The above value corresponds to the Levator Scapulae Muscle right algometric site
Statistical Analysis 11: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.050, Mixed Models Analysis — The above p value corresponds to the Deltoid Muscle left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.51 — The above value corresponds to the Deltoid Muscle left algometric site
Statistical Analysis 12: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.068, Mixed Models Analysis — The above p value corresponds to the Deltoid Muscle right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.41 — The above value corresponds to the Deltoid Muscle right algometric site
Statistical Analysis 13: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.049, Mixed Models Analysis — The above p value corresponds to the Tibialis Anterior Muscle left algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.59 — The above value corresponds to the Tibialis Anterior Muscle left algometric site
Statistical Analysis 14: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.004, Mixed Models Analysis — The above p value corresponds to the Tibialis Anterior Muscle right algometric site. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.73 — The above value corresponds to the Tibialis Anterior Muscle right algometric site
Statistical Analysis 15: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null hypothesis: The effect of applying ATM does not differ in reducing the pain sensitivity assessed by the Pain Pressure Threshold (PPT) measured with the pressure algometer (Commander Algometer) in patients with chronic neck pain from applying A-S (main hypothesis); Test type: Other; p = 0.297, Mixed Models Analysis — The above p value corresponds to the Mastoid Process left algometric site. The threshold for statistical significance was p < 0.05. The above value correspond to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.03, Standard Error of Mean 0.03 — The above values correspond to the Mastoid Process left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 16: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.855, Mixed Models Analysis — The above p value corresponds to the Mastoid Process right algometric site. The threshold for statistical significance was p < 0.05. The above value correspond to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.004, Standard Error of Mean 0.03 — The above values correspond to the Mastoid Process right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 17: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.594, Mixed Models Analysis — The above p value corresponds to the Bladder 10 (BL 10) left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.01, Standard Error of Mean 0.02 — The above values correspond to the Bladder 10 (BL 10) left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 18: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.929, Mixed Models Analysis — The above p value corresponds to the Bladder 10 (BL 10) right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.002, Standard Error of Mean 0.02 — The above values correspond to the Bladder 10 (BL 10) right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 19: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.725, Mixed Models Analysis — The above p value corresponds to the Zygapophyseal Joint left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.002, Standard Error of Mean 0.05 — The above values correspond to the Zygapophyseal Joint left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 20: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.725, Mixed Models Analysis — The above p value corresponds to the Zygapophyseal Joint right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.01, Standard Error of Mean 0.02 — The above values correspond to the Zygapophyseal Joint right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 21: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.398, Mixed Models Analysis — The above p value corresponds to the Upper Trapezius Muscle left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.02, Standard Error of Mean 0.03 — The above values correspond to the Upper Trapezius Muscle left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 22: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.186, Mixed Models Analysis — The above p value corresponds to the Mastoid Process right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.04, Standard Error of Mean 0.03 — The above values correspond to the Upper Trapezius Muscle right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 23: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.833, Mixed Models Analysis — The above p value corresponds to the Levator Scapulae Muscle left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.01, Standard Error of Mean 0.02 — The above values correspond to the Levator Scapulae Muscle left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 24: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.469, Mixed Models Analysis — The above p value corresponds to the Levator Scapulae Muscle right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.02, Standard Error of Mean 0.03 — The above values correspond to the Levator Scapulae Muscle right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 25: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.399, Mixed Models Analysis — The above p value corresponds to the Deltoid Muscle left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.02, Standard Error of Mean 0.03 — The above values correspond to the Deltoid Muscle left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 26: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.752, Mixed Models Analysis — The above p value corresponds to the Deltoid Muscle right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.01, Standard Error of Mean 0.02 — The above values correspond to the Deltoid Muscle right algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 27: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.002, Mixed Models Analysis — The above p value corresponds to the Tibialis Anterior Muscle left algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.07, Standard Error of Mean 0.02 — The above values correspond to the Tibialis Anterior Muscle left algometric site. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 28: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 1, analysis 15]; Test type: Other; p = 0.003, Mixed Models Analysis — The above p value corresponds to the Tibialis Anterior Muscle right algometric site. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.07, Standard Error of Mean 0.02 — The above values correspond to the Tibialis Anterior Muscle right algometric site. The above values correspond to the comparison which is between groups at baseline

2. Secondary Outcome: Cervical Range of Motion Measured by the 3D Inertial Motion Moover® Sensor by SENSOR Medica Technology in Motion (Guidonia Montecelio, Roma, Italia)
Description: The 3D Inertial Motion Moover® Sensor of the company SENSOR medica Technology in Motion (Guidonia Montecelio, Roma, Italia) was used to record cervical range of motion by evaluating cervical spine motion, acceleration and rotation. The sensor was positioned in the center of the patients' forehead on the frontal bone at the level of the glabella and was fastened around the head with the assistance of a strap. Patients were seated with their back straight and their chin parallel to the floor while looking at a target corresponding to their field of view. They were then asked to perform 3 cervical movements (left-right rotation, left-right lateral flexion, flexion-extension) for 3 times each with a pause at each final position. Throughout the process, the examiner's assistant stabilized the patient's trunk and shoulders with their hands and encouraged their constant continuing of each movement.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
Degrees
  Rotation Maximum (Baseline) | 58.22 (9.33) | 63.22 (9.46)
  Rotation Maximum (Endline) | 63.63 (12.1) | 63.77 (8.9)
  Rotation Average (Baseline) | 55.78 (10) | 60.62 (9.84)
  Rotation Average (Endline) | 60.7 (14.69) | 61.61 (9.52)
  Lateral Flexion Maximum (Baseline) | 28.26 (6.83) | 30.4 (6.55)
  Lateral Flexion Maximum (Endline) | 32.07 (7.28) | 31.4 (7.06)
  Lateral Flexion Average (Baseline) | 27.5 (6.67) | 29.5 (6.49)
  Lateral Flexion Average (Endline) | 31.07 (6.9) | 30.73 (7.02)
  Flexion Maximum (Baseline) | 50.31 (10.3) | 51.22 (10.25)
  Flexion Maximum (Endline) | 54.83 (10.46) | 52.67 (8.04)
  Flexion Average (Baseline) | 49.21 (10.77) | 49.36 (10.28)
  Flexion Average (Endline) | 53.66 (10.82) | 51.48 (8.05)
  Extention Maximum (Baseline) | 57.09 (12.31) | 58.26 (12.45)
  Extention Maximum (Endline) | 62.94 (14) | 60.91 (10.86)
  Extention Average (Baseline) | 56.07 (11.85) | 56.1 (12.52)
  Extention Average (Endline) | 61.55 (13.66) | 59.37 (10.91)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null hypothesis: The application of ATM does not affect the cervical range of motion (ROM) recorded with the Moover three-dimensional (3D) Inertial Motion sensor in patients with chronic neck pain (secondary hypothesis); Test type: Other; p = 0.002, Mixed Models Analysis — The above p value corresponds to the Rotation maximum. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 5.41 — The above value corresponds to the Rotation maximum
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.046, Mixed Models Analysis — The above p value corresponds to the Rotation average. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 4.92 — The above value corresponds to the Rotation average
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p value corresponds to the Lateral Flexion maximum. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 3.81 — The above value corresponds to the Lateral Flexion maximum
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.043, Mixed Models Analysis — The above p value corresponds to the Lateral Flexion average. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 3.57 — The above value corresponds to the Lateral Flexion average
Statistical Analysis 5: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.018, Mixed Models Analysis — The above p value corresponds to the Flexion maximum. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 4.52 — The above value corresponds to the Flexion maximum
Statistical Analysis 6: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.102, Mixed Models Analysis — The above p value corresponds to the Flexion average. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 4.45 — The above value corresponds to the Flexion average
Statistical Analysis 7: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.160, Mixed Models Analysis — The above p value corresponds to the Extension maximum. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 5.85 — The above value corresponds to the Extension maximum
Statistical Analysis 8: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.039, Mixed Models Analysis — The above p value corresponds to the Extension average. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 5.48 — The above value corresponds to the Extension average
Statistical Analysis 9: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null hypothesis: The effect of the application of ATM does not differ in the improvement of the cervical ROM recorded with the Moover three-dimensional (3D) Inertial Motion sensor in patients with chronic neck pain from the application of A-S (secondary hypothesis); Test type: Other; p = 0.001, Mixed Models Analysis — The above p-value corresponds to the Rotation maximum. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -5.00, Standard Error of Mean 1.51 — The above values correspond to the Rotation maximum. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 10: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.002, Mixed Models Analysis; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -5.00, Standard Error of Mean 1.51 — The above values correspond to the Rotation average. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 11: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.048, Mixed Models Analysis — The above p value corresponds to the Lateral Flexion maximum. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -4.84, Standard Error of Mean 1.60 — The above values correspond to the Lateral Flexion maximum. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 12: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.059, Mixed Models Analysis — The above p value corresponds to the Lateral Flexion average. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -2.00, Standard Error of Mean 1.06 — The above values correspond to the Lateral Flexion average. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 13: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.57, Mixed Models Analysis — The above p value corresponds to the Flexion maximum. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.92, Standard Error of Mean 1.62 — The above values correspond to the Flexion maximum. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 14: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.931, Mixed Models Analysis — The above p value corresponds to the Flexion average. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.14, Standard Error of Mean 1.65 — The above values correspond to the Flexion average. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 15: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.558, Mixed Models Analysis — The above p value corresponds to the Extension maximum. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -1.17, Standard Error of Mean 1.99 — The above values correspond to the Extension maximum . The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 16: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 2, analysis 9]; Test type: Other; p = 0.989, Mixed Models Analysis — The above p value corresponds to the Extension average. The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.03, Standard Error of Mean 1.96 — The above values correspond to the Extension average. The above values correspond to the comparison which is between groups at baseline

3. Secondary Outcome: Endurance of Deep Cervical Flexor Muscles of the Spine Measured by Chattanooga Stabilizer Pressure Biofeedback (PRESSURE BIOREACTION STABILIZER )
Description: The stabilizer assesses the endurance of deep flexor muscles of the spine using the Cranio-Cervical Flexion Test (CCF Test). The changing pressure will be recorded in an air-filled pressure cell, which is connected to a combined guide and plier. The sack is filled up with air until the 20 mmHg indication is shown. There are 5 levels of motion corresponding to a range of 20-30 mmHg of pressure (Level 1: 22 (decreased endurance), Level 2:24, Level 3: 26, Level 4: 28, Level 5:30 (increased endurance)) with a 30-second break in between. Contraction in each level lasts for 10 seconds. If the patient is unable to endure their position for this amount of time in each level, the test is terminated. The efficiency index is calculated as the quotient where the numerator records the pressure increase in the chamber and the denominator the number of repetitions. The maximum applied pressure sustained for a period of ten seconds is defined as the degree of activation.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
mmHg
  Baseline | 28.03 (3.07) | 27.68 (3.1)
  Endline | 29.4 (2.06) | 29.33 (1.86)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null hypothesis: The application of ATM does not affect the strength of deep neck flexor muscles as measured by the Chattanooga Stabilizer Pressure Biofeedback in patients with chronic pain in the cervical spine (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 1.37
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of applying ATM does not differ in improving the strength of deep neck flexor muscles measured by the Chattanooga Stabilizer Pressure Biofeedback in patients with chronic neck pain than applying A-S (secondary hypothesis); Test type: Other; p = 0.437, Mixed Models Analysis — The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.01, Standard Error of Mean 0.01 — The above values correspond to the comparison which is between groups at baseline

4. Secondary Outcome: Forced Vital Capacity (FVC) Measured by the Spirometer MIR Spirodoc
Description: For the evaluation of the respiratory function, a portable spirometer of the MIR company (MIR Spirodoc) was used. The process involved the measurement of Forced Vital Capacity (FVC). Each patient was given a sterilized nozzle. They were then asked to seal it with their lips and breathe normally through it while their nasal airway was blocked with the use of a clip. Patients inhaled slowly and deeply through the nozzle. Once their lungs were fully filled up with air, they were encouraged to exhale explosively for a minimum duration of 6 seconds.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
Liters
  Baseline | 3.79 (0.97) | 4.25 (1.17)
  Endline | 3.81 (0.93) | 4.31 (1.24)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the respiratory function assessed by the portable spirometer (MIR Spirodoc) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p = 0.919, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.02
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the improvement of the respiratory function in patients with chronic neck pain from the application of A-S (secondary hypothesis); Test type: Other; p = 0.010, Mixed Models Analysis — The above value corresponds to the comparison between groups at baseline. The threshold for statistical significance was p < 0.05; Dependence coefficients (β) = -0.05, Standard Error of Mean 0.02 — The above value corresponds to the comparison between groups at baseline

5. Secondary Outcome: Vital Capacity (VC) Measured by the Spirometer MIR Spirodoc
Description: For the evaluation of the respiratory function, a portable spirometer of the MIR company (MIR Spirodoc) was used. The process involved the measurement of Vital Capacity (VC).
  Each patient was given a sterilized nozzle. They were then asked to seal it with their lips and breathe normally through it while their nasal airway was blocked with the use of a clip. Patients inhaled slowly and deeply through the nozzle. Once their lungs were fully filled up with air, they were encouraged to exhale slowly and extensively until the lungs were fully emptied.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
Liters
  Baseline | 3.25 (0.93) | 3.67 (1.37)
  Endline | 3.34 (1) | 3.71 (1.3)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.659, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 0.09
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.05, Mixed Models Analysis — The above value correspond to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.04, Standard Error of Mean 0.02 — The above value correspond to the comparison which is between groups at baseline

6. Secondary Outcome: Maximum Voluntary Ventilation (MVV) Measured by the Spirometer MIR Spirodoc
Description: For the evaluation of the respiratory function, a portable spirometer of the MIR company (MIR Spirodoc) was used. The process involved the measurement of Maximum Voluntary Ventilation (MVV).
  Each patient was given a sterilized nozzle. They were then asked to seal it with their lips and breathe normally through it while their nasal airway was blocked with the use of a clip. This test contains a rhythmical and fast rotation of deep inhalations and exhalations until a distinctive auditory signal is sounded after 15 seconds.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: Liters/minutes
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
Liters/minutes
  Baseline | 101.88 (30.03) | 118.34 (38.12)
  Endline | 112.16 (34.6) | 122.82 (38.76)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.09, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 10.28
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.06, Standard Error of Mean 0.02 — The above value correspond to the comparison which is between groups at baseline

7. Secondary Outcome: Intensity and Quality of Pain Measured by the Short Form McGill Pain Questionnaire.
Description: The Short Form McGill Pain Questionnaire (SFMPQ) consists of 15 descriptors of pain sensation -11 sensory and 4 affective. The patient rates each description on a four-point intensity scale (0 - no pain, 1 - mild pain, 2 - moderate pain, and 3 - severe pain). The total score ranges from 0 to 45 points, the sensory subscale score from 0 to 33 points and the affective subscale score from 0 to 12 points. The higher the total score on the SFMPQ, the more the pain experience for the patient increases, indicating worse outcome. The Visual Analogue Scale (VAS) and the Present Pain Intensity (PPI) scale are included in the SFMPQ.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Sensory Score (Baseline) | 10.24 (6.73) | 9.84 (5.78)
  Sensory Score (Endline) | 4.69 (5) | 5.18 (5.45)
  Affective Score (Baseline) | 3.66 (3.77) | 3.04 (2.61)
  Affective Score (Endline) | 1.33 (2.12) | 1.47 (2.34)
  Total McGill Score (Baseline) | 13.89 (9.86) | 12.88 (7.76)
  Total McGill Score (Endline) | 6.02 (6.81) | 6.65 (7.42)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the pain in the cervical spine in terms of its intensity and quality, i.e., its sensory, emotional and behavioral dimensions using the McGill Pain Questionnaire-short form (SFMPQ) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Total McGill Score. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -7.87 — The above value corresponds to the Total McGill Score
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Sensory Score. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -5.55 — The above value corresponds to the Sensory Score
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Affective Score. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.33 — The above value corresponds to the Affective Score
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the reduction of pain in terms of its intensity and quality in patients with chronic neck pain from the application of A-S (secondary hypothesis); Test type: Other; p = 0.996, Mixed Models Analysis — The above p-value corresponds to the Total McGill score. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models. The above p-value corresponds to the comparison which is between groups at baseline; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.05 — The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 5: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 7, analysis 4]; Test type: Other; p = 0.968, Mixed Models Analysis — The above p-value corresponds to the Sensory Score. The threshold for statistical significance was p < 0.05; [statistical method as in outcome 7, analysis 4]; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.05 — The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 6: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 7, analysis 4]; Test type: Other; p = 0.854, Mixed Models Analysis — The above p-value corresponds to the Affective Score. The threshold for statistical significance was p < 0.05; [statistical method as in outcome 7, analysis 4]; Dependence coefficient (β) = 0.01, Standard Error of Mean 0.05 — The above values correspond to the comparison which is between groups at baseline

8. Secondary Outcome: Pain Intensity Measured by the Visual Analogue Scale
Description: The Visual Analogue Scale (VAS) measures pain intensity, asking the patient to rate their current or past level of pain by placing a mark on the line. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The following cut points have been recommended: no pain (0-0,4 cm), mild pain(0,5-4,4 cm), moderate pain (4,5-7,4 cm), and severe pain (7,5-10 cm). A higher score indicates higher pain intensity corresponding to a worse outcome.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Baseline | 4.36 (1.82) | 4.5 (2.18)
  Endline | 1.77 (1.71) | 2.25 (1.91)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Test type: Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.59
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Test type: Other; p = 0.952, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.03 — The above values correspond to the comparison which is between groups at baseline

9. Secondary Outcome: Present Pain Intesity Measured by the Present Pain Intensity Index.
Description: The Present Pain Intensity (PPI) is a six-point rating scale, which ranges from 0 to 5 (0=No pain, 1=Mild, 2 =Annoying, 3=Painful, 4=Horrible, 5=Unbearable). The descriptions are ranked according to increasing intensity so each of them can reflect a higher score. The higher point corresponds to worse outcome.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Baseline | 1.78 (0.7) | 1.82 (0.87)
  Endline | 0.72 (0.66) | 0.9 (0.7)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Test type: Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; Log transformation was used for the mixed linear models; Mean Difference (Net) = -1.06
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Test type: Other; p = 0.989, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.02 — The above values correspond to the comparison which is between groups at baseline

10. Secondary Outcome: Neck Disability Measured by the Neck Disability Index
Description: Neck Disability Index (NDI) consists of ten items, each of them corresponds to six answers from which the patient must choose only one. The lowest score for each item is zero which is assigned as no pain and no functional limitation and the maximum is five which refers to the worst pain and maximum limitation. Therefore, it is understandable that the total score ranges from zero to fifty, with values 0-4 (0%-8%) corresponding to no disability, 5-14 (10%-28%) to mild disability, 15-24 (30%-48%) to moderate disability, 25-34 (50%-68%) to severe and 35-50 (70%-100%) to absolute disability (higher scores mean a worse outcome).
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Baseline | 12.22 (5.76) | 11.92 (5.11)
  Endline | 6.62 (5.57) | 5.82 (5.03)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the functionality recorded with the Neck Disability Index (NDI) in patients with chronic pain in the cervical spine (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -5.6
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the improvement of functionality recorded with the Neck Disability Index (NDI) in patients with chronic neck pain from the application of A-S (secondary hypothesis); Test type: Other; p = 0.973, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.03 — The above value corresponds to the comparison which is between groups at baseline

11. Secondary Outcome: Anxiety and Depression Measured by the Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-report scale of 14 items, which are rated on a four-point scale numbered 0-3. It has two subscales, HADS_anxiety and HADS_depression, each of which contains seven items. The total score ranges from 0-21 for each subscale, where values 0-7 correspond to normal depression/anxiety, 8-10 to borderline abnormal depression/anxiety, and 11-21 to abnormal depression/anxiety (higher scores mean a worse outcome).
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Depression Sub-scale (Baseline) | 5.68 (3.63) | 4.86 (2.72)
  Depression Sub-scale (Endline) | 3.57 (3.19) | 3.41 (3.05)
  Anxiety Sub-scale (Baseline) | 8.67 (3.82) | 7.82 (3.69)
  Anxiety Sub-scale (Endline) | 6.62 (3.4) | 5.84 (3.76)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the anxiety and depression captured by the Hospital Anxiety & Depression Scale (HADS) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Depression subscale of HADS. The threshold for statistical significance was p < 0.05; Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.11 — The above value corresponds to the Depression subscale of HADS
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 11, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above value corresponds to the Anxiety subscale of HADS. The threshold for statistical significance was p < 0.05; Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.05 — The above value corresponds to the Anxiety subscale of HADS
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the reduction of anxiety and depression captured by the Hospital Anxiety & Depression Scale (HADS) in patients with chronic pain in the cervical spine from the application of A-S (secondary hypothesis); Test type: Other; p = 0.305, Mixed Models Analysis — The above p-value corresponds to the Depression subscale of HADS. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.04, Standard Error of Mean 0.04 — The above values correspond to the Depression subscale of HADS. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 11, analysis 3]; Test type: Other; p = 0.137, Mixed Models Analysis — The above p-value corresponds to the Anxiety subscale of HADS. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.05, Standard Error of Mean 0.03 — The above values correspond to the Anxiety subscale of HADS. The above values correspond to the comparison which is between groups at baseline

12. Secondary Outcome: Kinesiophobia Measured by the Tampa Scale Kinesiophobia
Description: The Tampa Scale Kinesiophobia (TSK) is a 17-item questionnaire with a score of 17-68.
  Four values correspond to each of the 17 questions: 1=Strongly disagree, 2=Disagree to some extent, 3=Agree to some extent, 4=Strongly agree, while the total score is obtained after reversing questions 4, 8, 12 and 16. If the latter amounts to 37 or less then it is associated with a low fear of movement, while on the contrary, 37 or more, with an increased one.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Baseline | 36.71 (7.58) | 35.01 (6.94)
  Endline | 32.89 (6.54) | 32.06 (6.53)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the kinesiophobia as measured by the Tampa Scale Kinesiophobia (TSK_GR) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -3.82
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ from the application of A-S in reducing kinesiophobia measured by the Tampa Scale Kinesiophobia (TSK_GR) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p = 0.151, Mixed Models Analysis — The threshold for statistical significance was p < 0.05. The above value corresponds to the comparison which is between groups at baseline; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.02, Standard Error of Mean 0.01 — The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement; Test type: Other; p = 0.021, McNemar — The threshold for statistical significance was p < 0.05

13. Secondary Outcome: Perception of Fear and Trying to Avoid Pain in Relation to Physical and Work Activities Measured by the Fear Avoidance Beliefs Questionnaire.
Description: The Fear Avoidance Beliefs Questionnaire (FABQ) is a self-referential questionnaire consisting of 16 questions, each of which is scored from zero to six. Therefore, the total score is 96 points. Higher scores correspond to strong perceptions of fear and avoiding pain, indicating a worse outcome. It consists of two subscales; the FABQ_physical (FABQ-P) composed of four questions and assessing the aforementioned parameters in relation to physical activities and the FABQ_work (FABQ-W), comprised of seven questions on the same perceptions at work, with scores ranging between 0-24 (15 or greater is considered a high score) and 0-42 (34 or greater is considered a high score with a higher probability of not returning to work) respectively. The remaining five questions aim to distract the patient.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  FABQ_Physical Subscale (Baseline) | 14.54 (5.6) | 12.91 (5.38)
  FABQ_Physical Subscale (Endline) | 10.3 (5.81) | 9.8 (5.47)
  FABQ_Work Subscale (Baseline) | 16.8 (8.9) | 14.05 (8.33)
  FABQ_Work Subscale (Endline) | 14.56 (8.8) | 10.57 (8.59)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the perception of the fear and the effort to avoid pain in relation to physical and work activities assessed by the Fear Avoidance Beliefs Questionnaire_Greek version (FABQ_GR) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p = 0.006, Mixed Models Analysis — The above p-value corresponds to the FABQ_physical subscale. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -4.24 — The above value corresponds to the FABQ_physical subscale
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.001, Mixed Models Analysis — The above p-value corresponds to the FABQ_work subscale. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.24 — The above value corresponds to the FABQ_work subscale
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the improvement of perception of fear and effort to avoid pain in relation to physical and work activities assessed by the Fear Avoidance Beliefs Questionnaire_Greek version (FABQ_GR) in patients with chronic neck pain from the application of A-S (secondary hypothesis); Test type: Other; p = 0.197, Mixed Models Analysis — The above p-value corresponds to the FABQ_work subscale. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.10, Standard Error of Mean 0.07 — The above values correspond to the FABQ_work subscale. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 13, analysis 3]; Test type: Other; p = 0.066, Mixed Models Analysis — The above p-value corresponds to the FABQ_physical subscale. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.07, Standard Error of Mean 0.04 — The above values correspond to the FABQ_physical subscale. The above values correspond to the comparison which is between groups at baseline

14. Secondary Outcome: Pain Catastrophizing Measured by the Pain Catastrophizing Scale.
Description: The Pain Catastrophizing Scale (PCS) scale is a 13-item instrument derived from the definitions of catastrophizing analyzed in the literature and from items from the catastrophizing subscale of the Coping Strategies Questionnaire (CSQ). Participants will be asked to recall past painful experiences and rate each of 13 thoughts or feelings on a five-point scale, where zero (0) corresponds to not at all and four (4) to constantly/all the time. The total score is calculated from the sum of the individual 13 question scores and ranges from 0 to 52. The Rumination subscale score ranges from 0 to 16 points, the Magnification subscale score from 0 to 12 points and the Helplessness subscale score from 0 to 24 points. Higher scores indicate a greater degree of pain catastrophizing meaning a worse outcome. A total score of >30 represents a clinically significant level of pain catastrophization, while a score of zero corresponds to no pain catastrophizing thoughts.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Rumination (Baseline) | 7.87 (4.62) | 7.64 (4.12)
  Rumination (Endline) | 5.85 (4.27) | 5.27 (4.7)
  Magnification (Baseline) | 4.21 (3.16) | 3.87 (2.49)
  Magnification (Endline) | 2.55 (2.64) | 2.41 (2.43)
  Helplessness (Baseline) | 9.01 (5.91) | 8.71 (5.3)
  Helplessness (Endline) | 5.62 (5.16) | 5.51 (4.98)
  PCS Total Score (Baseline) | 21.09 (12.28) | 20.22 (10.6)
  PCS Total Score (Endline) | 14.02 (10.93) | 13.2 (11.25)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the degree of pain catastrophizing recorded by the Pain Catastrophizing Scale (PCS) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Total PCS score. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -7.07 — The above value corresponds to the Total PCS score
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 14, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Rumination subscale of PCS. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -2.02 — The above value corresponds to the Rumination subscale of PCS
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 14, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Magnification subscale of PCS. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -1.66 — The above value corresponds to the Magnification subscale of PCS
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 14, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Helplessness subscale of PCS. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = -3.39 — The above value corresponds to the Helplessness subscale of PCS
Statistical Analysis 5: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ from the application of A-S in reducing pain catastrophizing recorded by the Pain Catastrophizing Scale (PCS) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p = 0.871, Mixed Models Analysis — The above p-value corresponds to the Total PCS score. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.01, Standard Error of Mean 0.05 — The above values correspond to the Total PCS score. The above values correspond to the comparison which is between groups at baseline; The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 6: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 14, analysis 5]; Test type: Other; p = 0.887, Mixed Models Analysis — The above p-value corresponds to the Rumination subscale of PCS. The above value correspond to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.01, Standard Error of Mean 0.06 — The above values correspond to the Rumination subscale of PCS. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 7: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 14, analysis 5]; Test type: Other; p = 0.879, Mixed Models Analysis — The above p-value corresponds to the Magnification subscale of PCS. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.01, Standard Error of Mean 0.05 — The above values correspond to the Magnification subscale of PCS. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 8: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 14, analysis 5]; Test type: Other; p = 0.961, Mixed Models Analysis — The above p-value corresponds to the Helplessness subscale of PCS. The above value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = 0.00, Standard Error of Mean 0.05 — The above values correspond to the Helplessness subscale of PCS. The above values correspond to the comparison which is between groups at baseline

15. Secondary Outcome: Quality of Life Measured by the Short Form 12 Health Survey.
Description: The Short Form (SF)-12 Health Survey is the short form of the SF-36 which contains 12 out of 36 questions. It assesses the parameters physical functioning (PF), physical and emotional role (role physical/RP, role emotional/RE) and mental health (MH), using two items. The parameters bodily pain (BP), general health (GH), social functioning (SF) and vitality (VT) are represented by a single item. All 12 items are used to measure the physical and mental component summary scores (PCS-12 and MCS-12). Scores in subscales range from 0 to 100 and higher scores are indicative of better mental and physical health status and better outcome. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Time Frame: Participants were assessed before (at baseline) and after (five weeks) the completion of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale
  Physical Component Summary Score (Baseline) | 44.98 (9.86) | 45.75 (7.54)
  Physical Component Summary Score (Endline) | 49.97 (7.47) | 50.41 (7.01)
  Mental Component Summary Score (Baseline) | 43.83 (9.46) | 46.89 (8.46)
  Mental Component Summary Score (Endline) | 52.16 (7.96) | 51.35 (5.98)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement; Null Hypothesis: The application of ATM does not affect the quality of life as measured by the Short Form 12-item Health Survey (SF-12) in patients with chronic neck pain (secondary hypothesis); Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Physical Component Summary/PCS subscale of SF-12. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 4.99 — The above value corresponds to the Physical Component Summary/PCS subscale of SF-12
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; [analysis description as in outcome 15, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — The above p-value corresponds to the Mental Component Summary/MCS subscale of SF-12. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Mean Difference (Net) = 8.33 — The above value corresponds to the Mental Component Summary/MCS subscale of SF-12
Statistical Analysis 3: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Null Hypothesis: The effect of the application of ATM does not differ in the improvement of quality of life measured by the Short Form 12-item Health Survey (SF-12) in patients with chronic pain in the cervical spine from the application of A-S (secondary hypothesis); Test type: Other; p = 0.564, Mixed Models Analysis — The above p-value corresponds to the Physical Component Summary/PCS of SF-12. The above p-value corresponds to the comparison which is between groups at baseline. The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -0.76, Standard Error of Mean 1.32 — The above values correspond to the Physical Component Summary/PCS subscale of SF-12. The above values correspond to the comparison which is between groups at baseline
Statistical Analysis 4: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; [analysis description as in outcome 15, analysis 3]; Test type: Other; p = 0.023, Mixed Models Analysis — The above p-value corresponds to Mental Component Summary/MCS of SF-12. The above p-value corresponds to the comparison which is between groups at baseline.The threshold for statistical significance was p < 0.05; The Log transformation was used for the mixed linear models; Dependence coefficient (β) = -3.05, Standard Error of Mean 1.34 — The above values correspond to the Mental Component Summary/MCS of SF-12. The above values correspond to the comparison which is between groups at baseline

16. Secondary Outcome: Global Perceived Effect Measured by the Global Perceived Effect Scale
Description: The Global Perceived Effect (GPE) cale was used to assess the perceived change of the subject's health condition. It asks the patient to rate how much their condition has worsened or improved relatively to another predetermined point in time (before the treatments). It is a numerical scale which consists of only one question with 5 possible answers. Values range between 1-5 with the higher score indicating worse outcome.
Time Frame: Participants were assessed after the completion of the interventions (five weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
Number analyzed (Participants) | 76 | 76
score on a scale | 1.49 (0.58) | 1.78 (0.64)
Statistical Analysis 1: Comparison: Feldenkrais Awareness Through Movement vs Acupuncture and Stretching; Test type: Other; p = 0.014, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05
Statistical Analysis 2: Comparison: Feldenkrais Awareness Through Movement; Test type: Other; Median Difference (Net) = 1
Statistical Analysis 3: Comparison: Acupuncture and Stretching; Test type: Other; Median Difference (Net) = 2

ADVERSE EVENTS:
Time Frame: Data was collected the period the intervention started and finished (5 weeks). However, more time was given in case of complications and adverse effects reported by the patients, which would be included in the analysis, assessed up to 10 weeks.
Arm/Group | Feldenkrais Awareness Through Movement | Acupuncture and Stretching
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76

LIMITATIONS AND CAVEATS:
There are several limitations. Firstly, the numerous exclusion criteria applied on the patients could affect the generalization of the results. Secondly, there is potential bias due to the lack of patients' and physiotherapists' blinding. Thirdly, the long-term efficacy of FM could not be evaluated because of the absence of a follow-up period. Another limitation is represented by the heterogeneity in the severity of the patients' symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT05870371/Prot_SAP_004.pdf
  • Informed Consent Form (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT05870371/ICF_005.pdf